CLINICAL TRIAL: NCT04491747
Title: Assessment of Factors That Affected Respiratory Parameters in Mucopolysaccharidoses Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Kılıç, Physiotherapist, Hacettepe University
Other Study IDs: GO 19/97
Record Dates: First submitted 2020-07-19; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Mucopolysaccharidoses
Keywords: Respiratory muscles; exercise test
MeSH Terms: conditions — Mucopolysaccharidoses | interventions — Functional Residual Capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: functional capacity — Six minute walk test used assessment of functional capacity.
  Other Names: Exercise capacity

SUMMARY:
Respiratory system affects in mucopolysaccharidosis (MPS) disease. Respiratory system symptoms are seen in almost every MPS patients and respiratory failure is one of the most common causes of death in this population. The aim of the study was to evaluate respiratory muscle strength and endurance, cough effectiveness and functional capacity in MPS patients and to defined the factors that affected the respiratory problem in this.

DETAILED DESCRIPTION:
This study was participated MPS patients. Patients' pulmonary function test, functional capacity, respiratory muscle strength and endurance, peak cough flow was assessed and recorded.

Pulmonary function test was assessed with spirometry, functional capacity was evaluated with 3-minute step test and six minute walk test (MWT). Respiratory muscle strength was evaluated mouth pressure measurement (MIP- maximal inspiratory pressure and MEP- maximal expiratory pressure) and Sniff nasal inspiratory pressure (SNIP). Respiratory muscle endurance was assessed Powerbreathe. And cough effectiveness was evaluated peak cough flow.

ELIGIBILITY:
Inclusion Criteria:

* People who diagnosed Mucopolysaccharidoses disease in Hacettepe University.
* Cooperation

Exclusion Criteria:

* Patients who were not walking ability.

Ages: 7 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: People who diagnosed Mucopolysaccharidoses disease in Hacettepe University were recruited the study.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
functional capacity | 15 minutes
  Six minute walk test: Distance walked in six minute was recorded
3 minute step test | 5 minutes
  number of completed step in 3 minute was recorded
Respiratory muscle strength assessment | 15 minutes
  Respiratory muscle strength was evaluated by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) and sniff nasal inspiratory pressure(SNIP). Also dynamic inspiratory muscle strength was evaluated Powerbreathe K5 device.
Respiratory muscle endurance | 10 minutes
  Pressure time unit: A constant load test was used to evaluate respiratory muscle endurance. Using a PowerBreathe device (HaB International Ltd., Southam, UK), the participants were asked to breathe maintaining a constant threshold (60% of MIP) until task failure, and the test duration was recorded. Results were obtained by multiplying the set pressure by the test duration
Pulmonary functions | 15 minutes
  FVC (Forced vital capacity) assessment via spirometry
Pulmonary functions | 15 minutes
  FEV 1(forced expiratory volume in first second) assessment via spirometry
Pulmonary functions | 15 minutes
  PEF (peak expiratory flow) assessment via spirometry
MVV (Maximal ventilatory assesssment) | 5 minutes
  Maximize ventilation by inhaling and exhaling as quickly and deeply as possible for 15 s via spirometry
cough effectiveness | 5 minutes
  cough effectiveness assessment was evaluated peak cough flow meter.

SECONDARY OUTCOMES:
heart rate | 6 minutes
  difference pre and post test heart beat number
oxygen saturation | 6 minutes
  difference pre and post test percentage of oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Dogru- Ersoz, Professor, Study Director — Hacettepe University; Naciye Vardar- Yagli, PhD, Study Chair — Hacettepe University; Dilber Ademhan- Tural, MD, Study Chair — Hacettepe University; Nural Kiper, Professor, Study Chair — Hacettepe University; Ugur Ozcelik, Professor, Study Chair — Hacettepe University; Ebru Yalcin, Professor, Study Chair — Hacettepe University; Deniz Inal-Ince, Professor, Study Chair — Hacettepe University; Melda Saglam, PhD, Study Chair — Hacettepe University; Serap Sivri, Professor, Study Chair — Hacettepe University; Aysegul Tokatlı, Professor, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)